CLINICAL TRIAL: NCT00488943
Title: Follow-up After Endovascular Repair of Abdominal Aortic Aneurysm
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: H53537-26003
Record Dates: First submitted 2007-06-18; First posted 2007-06-20 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Stent-Graft; AAA; Abdominal Aortic Anuerysm; Zenith; Endovascular; Treatment with Zenith Aortic Stent-Graft for repair Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: AAA Endovascular Bifurcated Stent-Graft — Treatment of Abdominal Aortic Aneurysm with a Zenith Endovascular Bifurcated Stent-Graft.
  Other Names: Zenith AAA Endovascular Stent-Graft (Cook, Inc.)

SUMMARY:
To collect and analyze clinical follow-up data which can be used to assess the safety, efficacy, and durability of endovascular AAA repair with Zenith and Chuter-Gianturco stent-grafts.

DETAILED DESCRIPTION:
We propose to analyze the data collected for clinical purposes in 453 patients who already underwent endovascular AAA repair at UCSF and SFVA, and others who will undergo this operation in the future. Most of these patients have now passed the 2-year follow-up required by the original protocol, all continue to be followed for clinical purposes, using the same studies, the same data forms and the same schedule as before, because studies of various devices of this type have shown that the potential for late problems requires continuing scrutiny of stent-graft structure and function, as a basis for timely re-intervention.

ELIGIBILITY:
Inclusion Criteria:

* AAA with diameter > 4 cm or AAA with a history of growth > 0.5 cm per year
* treatment of AAA with Zenith Stent-Graft

Exclusion Criteria:

* Pregnant
* Life expectancy less than two years
* Less than 18 years of age
* Unwilling to comply with clinical follow-up schedule
* Inability or refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Abdominal Aortic Aneurysms treated with Zenith Stent-Graft
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2005-01 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2024-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy AM Chuter, MD, Principal Investigator — Professor of Surgery; Joseph H Rapp, MD, Principal Investigator — Professor of Surgery; Linda M Reilly, MD, Principal Investigator — Professor of Surgery
Locations (2):
- United States (2):
  - Division of Vascular Surgery, SFVAMC, San Francisco, California
  - Division of Vascular Surgery, UCSF, San Francisco, California

REFERENCES:
- [Background] Lee WA, Carter JW, Upchurch G, Seeger JM, Huber TS. Perioperative outcomes after open and endovascular repair of intact abdominal aortic aneurysms in the United States during 2001. J Vasc Surg. 2004 Mar;39(3):491-6. doi: 10.1016/j.jvs.2003.12.001. PMID 14981436
- [Background] Jacobs TS, Won J, Gravereaux EC, Faries PL, Morrissey N, Teodorescu VJ, Hollier LH, Marin ML. Mechanical failure of prosthetic human implants: a 10-year experience with aortic stent graft devices. J Vasc Surg. 2003 Jan;37(1):16-26. doi: 10.1067/mva.2003.58. PMID 12514573
- [Background] Beebe HG, Cronenwett JL, Katzen BT, Brewster DC, Green RM; Vanguard Endograft Trial Investigators. Results of an aortic endograft trial: impact of device failure beyond 12 months. J Vasc Surg. 2001 Feb;33(2 Suppl):S55-63. doi: 10.1067/mva.2001.111663. PMID 11174813
- [Background] Bertges DJ, Chow K, Wyers MC, Landsittel D, Frydrych AV, Stavropoulos W, Tan WA, Rhee RY, Fillinger MF, Fairman RM, Makaroun MS. Abdominal aortic aneurysm size regression after endovascular repair is endograft dependent. J Vasc Surg. 2003 Apr;37(4):716-23. doi: 10.1067/mva.2003.212. PMID 12663968